CLINICAL TRIAL: NCT05958043
Title: Performance of CAD/CAM Milled and 3D-printed Full-arch Implant-supported Provisionals Restorations: A Randomized Controlled Clinical Trial
Brief Title: Performance of CAD/CAM Milled and 3D-printed Full-arch Implant-supported Provisionals Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Gómez Polo, Associate Professor of conservative dentistry and prosthodontics, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22/170-EC_P
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2023-07

CONDITIONS: Edentulous Jaw; Dental Prosthesis Complication; Dental Prosthesis Failure
Keywords: CAD/CAM; 3D-Printed; Full-arch provisional
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D-printed group (Experimental): The patients randomized to the 3D-printed group will receive a 3D-printed full arch implant-supported provisional restoration.
  Interventions: Device: 3D- printed Full-arch Implant-supported Provisionals Restorations
- CAD/CAM- milled group (Other): The patients randomized to the CAD/CAM-milled group will receive a PMMA-milled full-arch implant-supported provisional restoration.
  Interventions: Device: CAD/CAM-milled Full-arch Implant-supported Provisionals Restorations

INTERVENTIONS:
Device: 3D- printed Full-arch Implant-supported Provisionals Restorations — The full-arch provisional restorations will be placed on dental implants that should be positioned to allow for the fabrication of a prosthesis that spans at least 12 units (from the right first molar to the left first molar, accepting distal extensions). Before completing the essential clinical data registration to produce an individual patient-oriented prosthesis, trans-epithelial abutments will be put at the torque the manufacturer recommends (30-35 Ncm typically), according to the appropriate gingival height.
  At visit three, the full-arch provisional will be screwed in using the manufacturer's specified torque (15 Ncm typically). For 12 to 15 weeks (about three months), the patient will be in the preliminary phase, during which time data will be gathered. Once the stipulated time has elapsed, the definitive prosthesis in monolithic zirconia prosthesis will be placed.
  Arms: 3D-printed group
Device: CAD/CAM-milled Full-arch Implant-supported Provisionals Restorations — The full-arch provisional restorations will be placed on dental implants that should be positioned to allow for the fabrication of a prosthesis that spans at least 12 units (from the right first molar to the left first molar, accepting distal extensions). Before completing the essential clinical data registration to produce an individual patient-oriented prosthesis, trans-epithelial abutments will be put at the torque the manufacturer recommends (30-35 Ncm typically), according to the appropriate gingival height.
  At visit three, the full-arch provisional will be screwed in using the manufacturer's specified torque (15 Ncm typically). For 12 to 15 weeks (about three months), the patient will be in the preliminary phase, during which time data will be gathered. Once the stipulated time has elapsed, the definitive prosthesis in monolithic zirconia prosthesis will be placed.
  Arms: CAD/CAM- milled group

SUMMARY:
This clinical trial aims to compare the performance of CAD/CAM-milled and 3D-printed full-arch implant-supported provisional restorations in patients at the Advanced Implant Prosthetics Clinic of the Complutense University of Madrid, of both sexes, over 18 years of age, edentulous upper, lower or both, whose treatment plan is at least a fixed implant-supported rehabilitation of the complete arch. The main question it aims to answer is if there are differences in the mechanical behavior and optical properties of the materials used as provisional materials in full-arch restorations on implants fabricated by CAD/CAM technology through machining or 3D printing.

Participants will:

- Receive milled (control material: PMMA; Multilayer PMMA block, HUGE; Shandong Huge Dental Material Corporation) or printed (test material: 3D impression resin; VarseoSmile Temp, Bego Bremer Goldschägerei Wilh. Herbst GmbH & Co. KG, Bremen) and they will be in provisional phase for 3 months doing daily life.

Researchers will compare PMMA (Multilayer PMMA block, HUGE; Shandong Huge Dental Material Corporation) and the printed-resin (3D impression resin; VarseoSmile Temp, Bego Bremer Goldschägerei Wilh. Herbst GmbH & Co. KG, Bremen) to see:

* Mechanical behavior and the absence of complications, fracture of the structure, material jumping or wear, loosening, or detachment.
* Optical properties, initial color, and degradation of the materials used

DETAILED DESCRIPTION:
BACKGROUND

Since the discovery of osseointegration by Professor Branemark, dental implants have been introduced into clinical practice and are currently one of the most demanded treatments, being considered the first choice for the rehabilitation of patients with partial or total edentulism. Of all of them, the rehabilitation of the completely edentulous patient is one of the greatest challenges for the professional, since it requires meticulous planning to restore the patient's function and improve esthetics.

In this regard, the introduction of CAD/CAM technology has been a major breakthrough since it allows, as its name suggests, computer assistance in the design and fabrication phase. Its inclusion in the design phase facilitates this process and communication between the clinician and the laboratory with the design file, which could be re-fabricated if there are any complications. P or its use at the manufacturing stage decreases the influence of the laboratory technician's skill and allows the use of new materials. To date, these new materials have been manufactured by milling from a solid disk, the most commonly used materials being polymethylmethacrylate (PMMA) and polyoxymethylene (POM).

In recent years, the industry has focused its efforts on manufacturing by additive technology, by 3D printing, which has different advantages compared to subtractive technology or milling; such as, for example, the greater use of the material or the reduced limitations when manufacturing geometries where milling cannot reach. Gradually, new materials for 3D printing are appearing, with more applications, being already possible the fabrication of models, removable prostheses, gingival masks, unloading splints, and long-lasting temporary prostheses, or surgical guides. Recently, a new material has appeared, whose properties could be comparable to those of the materials used today as temporaries, mainly polymethylmethacrylate (PMMA), which is made by milling from solid blocks.

JUSTIFICATION

The emergence of new biocompatible 3D printing materials- indicated even for definitive restorations, with mechanical properties similar to the materials currently used as temporary materials- raises the use of this fabrication technique for long-lasting temporary materials.

HYPOTHESIS

Null hypothesis (H0): There are no differences in the mechanical behavior and optical properties of the materials used as provisional material in full-arch restorations on implants manufactured by CAD/CAM technology by machining or 3D printing.

Alternative hypothesis (H1): There are differences in the mechanical behavior and optical properties of the materials used as provisional materials in full-arch restorations on implants fabricated by CAD/CAM technology through machining or 3D printing.

OBJECTIVES

General Objective:

To compare the mechanical behavior and optical properties of the materials used as provisional material in full-arch restorations on implants manufactured by CAD/CAM technology, by machining or 3D printing.

Specific Objectives:

* To analyze the mechanical behavior and the absence of complications, fracture of the structure, material jumping or wear, loosening or debonding of the materials used as provisional material in full-arch restorations on implants manufactured by CAD/CAM technology, by machining or 3D printing.
* To analyze the optical properties, initial color, and degradation of the materials used as provisional material in full-arch restorations on implants manufactured by CAD/CAM technology, by machining or 3D printing.

MATERIAL AND METHODS

The research protocol was reviewed and approved by the Hospital Clínico San Carlos ethics committee, which served the Faculty of Dentistry of the Complutense University of Madrid (22/170- EC_P).

Study design:

Prospective parallel-group randomized controlled clinical study following CONSORT guidelines.

Reference and study population:

The study population will consist of patients seen at the Advanced Implant Prosthetics Clinic of the Complutense University of Madrid, of both sexes, over 18 years of age, edentulous upper, lower, or both jaws, whose treatment plan is at least a full-arch implant-supported fixed restoration (at least from right first molar to left first molar) and who meet all the inclusion criteria but none of the exclusion criteria.

Once the informed consent has been read and explained, and any possible doubts regarding the treatment and the study have been resolved, patients must give their written informed consent to participate in the study prior to any study-related procedure.

Data collection and information sources:

The data required for this study will be collected by a single investigator, using a case report form (CRF) for all patients from whom we obtain informed consent is obtained. First name initials will be used to code and track information for each patient. Also, will be coded numerically for each interim as the subject of study during the conduct of the study.

The patient will not know what temporary material the temporary restoration is made of.

* Demographic data: Subject demographics, including age, sex, and smoking habit, will be documented at the screening visit. Smoking habits will be classified in:

  * Non-smoker.
  * Smoker:

    * Mild: 5 or fewer cigarettes a day or one cigar a day.
    * Moderate: 6 to 15 cigarettes per day.
    * Severe: more than 16 cigarettes per day on average or more than one cigar per day (note: exclusion criteria).
    * Electronic cigarette consumer.
* General health status and dental history: General health status and dental history will be obtained at the screening visit. The investigator will assess relevant medical history and current medical conditions, based on available information, and classify the patient according to the ASA physical status classification system (18). Information may be obtained from the subject's general practitioner or from oral communication with the subject.

General health subjects' will be classified into:

* ASA I: Normal healthy patient (no acute or chronic diseases), healthy, non-smoker, no or minimal alcohol consumption. BMI and normal percentile for age.
* ASA II: Patient with mild systemic disease (only without substantial functional limitations), including current smokers, social alcohol drinkers, pregnant and/or patients with obesity, well-controlled DM/HTA, and mild pulmonary disease.
* ASA III: A patient with severe systemic disease (note: exclusion criteria). o ASA IV: A patient with a severe systemic illness that poses a constant threat to life (note: exclusion criteria).
* ASA V: A dying patient who is not expected to survive surgery (note: exclusion criteria).

Dental history:

* Indicate reasons for dental losses or extractions of the jaw to be rehabilitated.
* Indicate the presence of severe bruxing or clenching habits (note: exclusion criteria).

Diagnostic imaging: A panoramic radiograph should be available at the screening visit to evaluate anatomical structures and dentition. E n case it is available, it will be used for treatment planning. The panoramic radiograph may be taken during the screening visit or be available from an earlier date within 6 months.

STATISTICAL ANALYSIS

The variables will be recorded in a Microsoft Excel spreadsheet and analyzed by professional statisticians using specific software (IBM SPSS Statistics, v25 for Windows; IBM Corp.). The statistical analysis will include tests to determine whether the distribution of the data complies with normality principles (Shapiro- Wilk test) and then perform the inferential analysis. For the analysis of the optical behavior, a t-student for related samples will be used, and for the analysis of the mechanical behavior data, a repeated measures analysis of variance (ANOVA) will be used. Once it has been checked in an a priori test whether there are statistically significant differences, if they appear, a posteriori test (Tuckey test) will be performed to determine between which groups they occur.

STUDY LIMITATIONS

One of the study's main limitations is the recruitment of patients since completely edentulous patients are increasingly less prevalent in our society. In addition, they must be in good health and have good bone availability, which makes them susceptible to inclusion in the study. On the other hand, planning for this type of patient is laborious and often requires previous treatments (such as extractions or basic periodontal treatment) that lengthen the treatment time.

CHRONOGRAM / WORK PLAN

* January 2022 - February 2022: Study design, obtain ethics committee approval.
* March 2022 -April 2025: Patient treatment and data collection.
* April 2025 - July 2025: Data analysis and statistical study.
* September 2025 - December 2025: Report writing and possible manuscripts for publication in indexed journals.

PROTOCOL AMENDMENTS

Protocol changes will be kept to a minimum. Only those changes that are deemed essential to the successful completion of the protocol will be considered.

PUBLICATION RIGHTS

Analysis of data will be conducted by Data Management. The final manuscript will be prepared by the principal investigator in conjunction with sub-investigators and submitted for publication. Additionally, the results of the study will be entered on clinicaltrials.gov.

If it's decided on the future sharing of the IPD the following data will be shared and available:

* Participant's data that underlie the results reported in this article, after deidentification (text, tables, figures).
* The data and protocols may be only available to investigators and researchers who provide a methodologically sound proposal for individual participant data meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age.
* Healthy patients; ASA I or ASA II.
* Maxillary, mandibular, or both maxillary edentulous patients whose prosthetic treatment plan is a full-arch implant-supported fixed prosthesis.
* Patients must have voluntarily signed informed consent, be willing and able to attend scheduled follow-up visits, and agree to have coded data collected and analyzed.

Exclusion Criteria:

* Any contraindications for oral surgical procedures.
* Smokers classified as "heavy smokers" above 10 cigarettes per day (or more than 1 cigar per day) or smokers of chewing tobacco.
* Subjects with drug or alcohol abuse.
* Severe bruxing habits.
* Conditions or circumstances that, in the opinion of the investigator, would preclude completion of participation in the study or interfere with the analysis of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Mechanical behavior of 3D-resin and PMMA-milled materials used as provisional materials in full-arch restorations on implants fabricated by CAD/CAM technology. | 2 years
  The mechanical behavior will be evaluated on the basis of the occurrence of some mechanical complications. The mechanical complications to be evaluated will be classified by visual inspection in clinical examination as follows:
  * Appearance of material skips, minor fractures and/or chipping
  * Appearance of major fractures defined as an appearance of a broken structure that restrain the use of the devise.
Optical properties of 3D-resin and PMMA-milled materials used as provisional materials in full-arch restorations on implants fabricated by CAD/CAM technology. | 2 years
  The optical properties of the material will be based on the initial color of the material and its degradation from color acquisition using a Vita Easyshade® compact spectrophotometer (Vita, Zahnfabrik - Germany). Five measurements of tooth 1.1 or 4.1 depending on the maxilla will be taken on the day of provisional placement and after three months, the system code of the VITA classical and 3D Master shade guides will also be recorded. In addition, the coordinates of the CIELAB chromatic notation system will be recorded with which the brightness (L), chroma (C) and hue (h) and the differences in brightness (∆L) , chroma differences (∆C) and hue differences (∆H) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Gómez Polo, DDS, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- School of Dentistry, Complutense University. Pza Ramón y Cajal s/n., Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
If it is decided on the future sharing of the IPD the following data will be shared and available:
  * Participant's data that underlie the results reported in this article, after deidentification (text, tables, figures).
  * Other documents that would be available: Study protocol. The data and protocols may be only available to investigators and researchers who provide a methodologically sound proposal for individual participant data meta-analysis.
  The data would be available beginning 6 months and ending 5 years following article publication and it may be shared after a proposal is directed. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: the following data will be shared and available:
  * Participant's data that underlie the results reported in this article, after deidentification (text, tables, figures).
  * Other documents that would be available: Study protocol. The data and protocols may be only available to investigators and researchers who provide a methodologically sound proposal for individual participant data meta-analysis.
  The data would be available beginning 6 months and ending 5 years following article publication and it may be shared after a proposal is directed.
Access Criteria: To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] BRANEMARK PI, BREINE U. FORMATION OF BONE MARROW IN ISOLATED SEGMENT OF RIB PERIOSTEUM IN RABBIT AND DOG. Blut. 1964 Oct;10:236-52. doi: 10.1007/BF01630647. No abstract available. PMID 14290059
- [Background] Derksen W, Tahmaseb A, Wismeijer D. A Randomized Clinical Trial comparing the clinical fit of CAD/CAM monolithic zirconia Fixed Dental Prostheses (FDP) on ti-base abutments based on digital or conventional impression techniques. One year follow-up. Int J Prosthodont. 2021 November/December;34(6):733-743. doi: 10.11607/ijp.7074. Epub 2021 Mar 3. PMID 33662051
- [Background] Hensel F, Koenig A, Doerfler HM, Fuchs F, Rosentritt M, Hahnel S. CAD/CAM Resin-Based Composites for Use in Long-Term Temporary Fixed Dental Prostheses. Polymers (Basel). 2021 Oct 9;13(20):3469. doi: 10.3390/polym13203469. PMID 34685228
- [Background] Diez-Quijano C, Azevedo L, Antonaya-Martin JL, Del Rio-Highsmith J, Gomez-Polo M. Evaluation of the clinical behavior of 2 different materials for implant-supported interim fixed partial prostheses: A randomized clinical trial. J Prosthet Dent. 2020 Sep;124(3):351-356. doi: 10.1016/j.prosdent.2019.09.021. Epub 2019 Dec 4. PMID 31810613
- [Background] Mayer J, Reymus M, Wiedenmann F, Edelhoff D, Hickel R, Stawarczyk B. Temporary 3D printed fixed dental prosthesis materials: Impact of post printing cleaning methods on degree of conversion as well as surface and mechanical properties. Int J Prosthodont. 2021 November/December;34(6):784-795. doi: 10.11607/ijp.7048. Epub 2021 Feb 12. PMID 33616559
- [Background] Molinero-Mourelle P, Canals S, Gomez-Polo M, Sola-Ruiz MF, Del Rio Highsmith J, Vinuela AC. Polylactic Acid as a Material for Three-Dimensional Printing of Provisional Restorations. Int J Prosthodont. 2018 Jul/Aug;31(4):349-350. doi: 10.11607/ijp.5709. PMID 29953566
- [Background] Shin SH, Kwon JS, Shim JS, Kim JE. Evaluating the Three-Dimensional Printing Accuracy of Partial-Arch Models According to Outer Wall Thickness: An In Vitro Study. Materials (Basel). 2021 Nov 9;14(22):6734. doi: 10.3390/ma14226734. PMID 34832136
- [Background] Shin SH, Doh RM, Lim JH, Kwon JS, Shim JS, Kim JE. Evaluation of Dimensional Changes According to Aging Period and Postcuring Time of 3D-Printed Denture Base Prostheses: An In Vitro Study. Materials (Basel). 2021 Oct 18;14(20):6185. doi: 10.3390/ma14206185. PMID 34683773
- [Background] Srinivasan M, Kalberer N, Fankhauser N, Naharro M, Maniewicz S, Muller F. CAD-CAM complete removable dental prostheses: A double-blind, randomized, crossover clinical trial evaluating milled and 3D-printed dentures. J Dent. 2021 Dec;115:103842. doi: 10.1016/j.jdent.2021.103842. Epub 2021 Oct 9. PMID 34637889
- [Background] Tangpothitham S, Pongprueksa P, Inokoshi M, Mitrirattanakul S. Effect of post-polymerization with autoclaving treatment on monomer elution and mechanical properties of 3D-printing acrylic resin for splint fabrication. J Mech Behav Biomed Mater. 2022 Feb;126:105015. doi: 10.1016/j.jmbbm.2021.105015. Epub 2021 Nov 29. PMID 34896766
- [Background] Henderson JY, Korioth TVP, Tantbirojn D, Versluis A. Failure load of milled, 3D-printed, and conventional chairside-dispensed interim 3-unit fixed dental prostheses. J Prosthet Dent. 2022 Feb;127(2):275.e1-275.e7. doi: 10.1016/j.prosdent.2021.11.005. Epub 2021 Dec 10. PMID 34895902
- [Background] Crenn MJ, Rohman G, Fromentin O, Benoit A. Polylactic acid as a biocompatible polymer for three-dimensional printing of interim prosthesis: Mechanical characterization. Dent Mater J. 2022 Feb 1;41(1):110-116. doi: 10.4012/dmj.2021-151. Epub 2021 Dec 4. PMID 34866117
- [Background] Yang JW, Liu Q, Yue ZG, Hou JX, Afrashtehfar KI. Digital Workflow for Full-Arch Immediate Implant Placement Using a Stackable Surgical Guide Fabricated Using SLM Technology. J Prosthodont. 2021 Oct;30(8):645-650. doi: 10.1111/jopr.13375. Epub 2021 May 26. PMID 33938077
- [Background] Angelara K, Bratos M, Sorensen JA. Comparison of strength of milled and conventionally processed PMMA complete-arch implant-supported immediate interim fixed dental prostheses. J Prosthet Dent. 2023 Jan;129(1):221-227. doi: 10.1016/j.prosdent.2021.04.025. Epub 2021 Jun 20. PMID 34158174
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Browning WD, Contreras-Bulnes R, Brackett MG, Brackett WW. Color differences: polymerized composite and corresponding Vitapan Classical shade tab. J Dent. 2009;37 Suppl 1:e34-9. doi: 10.1016/j.jdent.2009.05.008. Epub 2009 May 18. PMID 19500895
- See also: World Health Organization. WHO Framework Convention on Tobacco Control — https://apps.who.int/iris/handle/10665/42811
- See also: Study Randomizer [App/Ethernet]. Wageningen. 2017 — https://www.studyrandomizer.com